CLINICAL TRIAL: NCT02670525
Title: Matched Targeted Therapy (MTT) Recommendation for Patients With Recurrent, Refractory, or High Risk Leukemias and Myelodysplastic Syndrome
Brief Title: Matched Targeted Therapy For High-Risk Leukemias and Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yana Pikman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-384
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Recurrent, Refractory, or High Risk Leukemias; Matched Targeted Therapy
Keywords: Recurrent, Refractory, or High Risk Leukemias; Matched targeted therapy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relapsed/Refractory Leukemia (Experimental): Cohort 1: Relapsed/Refractory Leukemia
  * Acute lymphoblastic leukemia (ALL), first or greater relapse
  * Acute myeloid leukemia (AML), first or greater relapse
  * Leukemia refractory to induction chemotherapy
  * Other recurrent leukemia
  * Myelodysplastic syndrome (MDS), first or greater relapse, or refractory to initial therapy
  After the screening procedures confirms patient eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Interventions: Genetic: Leukemia Profiling
- New Diagnosis (Experimental): Cohort 2: New Diagnosis
  * Acute myeloid leukemia (AML), new diagnosis (excluding acute promyelocytic leukemia (APL))
  * New diagnosis infant mixed-lineage leukemia (MLL)-rearranged ALL or low hypodiploid (<40 chromosomes) ALL
  * Rare leukemia- e.g., juvenile myelomonocytic leukemia (JMML), leukemia of ambiguous lineage
  * Secondary leukemia
  * Myelodysplastic syndrome (MDS) not eligible for stem cell transplant
  After the screening procedures confirms eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Interventions: Genetic: Leukemia Profiling

INTERVENTIONS:
Genetic: Leukemia Profiling — Genetic profiling of leukemia cells will be performed and analyzed by an expert panel. Matched targeted therapy recommendation based on profiling results will be made if available. The recommendation, if available, will be communicated to the primary oncologist.

SUMMARY:
This research study is seeking to gain new knowledge about Recurrent, Refractory, or High Risk Leukemias in children and young adults.

This study is evaluating the use of specialized testing called leukemia profiling. Once the profiling is performed, the results are evaluated by an expert panel of physicians, scientists and pharmacists. This may result in a recommendation for a specific cancer therapy or a clinical trial called matched targeted therapy (MTT). The results of the leukemia profiling and, if applicable, the MTT recommendation will be communicated to the participant's primary oncologist.

DETAILED DESCRIPTION:
Our tissues and organs are made up of cells. Cancer occurs when the molecules that normally control cell growth are damaged. The damage results in unchecked cell growth which causes a tumor, a collection of cancer cells. The damage is referred to as an alteration. There are different types of cancer-causing alterations. Genes are the part of cells that contain the instructions which tell our cells how to make the right proteins to grow and work. Genes are composed of Deoxyribonucleic Acid (DNA) letters that spell out these instructions.

By participating in this study, the participant's leukemia cells will be tested for cancer causing alterations. This testing is called leukemia profiling. The leukemia profiling will be performed using bone marrow or blood that has already been obtained during a clinical test. Alternately, the profiling may be done on leukemia cells that are planned to be obtained as part of routine clinical care.

This study will determine whether it is possible to use profiling results to determine a matched targeted therapy for patients with leukemia. It will describe the range of mutations found in patients with leukemia with this type of profiling, and describe the clinical outcomes of patients who receive a matched targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Birth to ≤ 30 years at study entry
* Diagnosis: Patients will be enrolled in one of the two cohorts based on diagnosis:

Cohort 1: Relapsed/refractory leukemia

* Acute lymphoblastic leukemia (ALL), first or greater relapse
* Acute myeloid leukemia (AML), first or greater relapse
* Leukemia refractory to induction chemotherapy
* Other recurrent leukemia
* Myelodysplastic syndrome (MDS), first or greater relapse, or refractory to initial therapy

Cohort 2: New diagnosis

* Acute myeloid leukemia (AML), new diagnosis
* New diagnosis infant mixed-lineage leukemia (MLL)-rearranged ALL or low hypodiploid (<40 chromosomes) ALL
* Rare leukemia- e.g., juvenile myelomonocytic leukemia (JMML), leukemia of ambiguous lineage
* Secondary leukemia
* Myelodysplastic syndrome (MDS) not eligible for stem cell transplant

Pathologic Criteria

* Histologic confirmation of leukemia at the time of diagnosis or recurrence

Specimen Samples

* Sufficient leukemia specimen available for profiling from diagnosis or recurrence OR bone marrow aspirate/blood draw/pheresis/other fresh sample of patient leukemia cells planned for clinical care anticipated to allow collection of minimum specimen for testing.

Exclusion Criteria:

* Insufficient leukemia specimen available for profiling from diagnosis or recurrence; or bone marrow evaluation/blood draw/other leukemia cell sample NOT planned to be obtained for clinical care; or peripheral blast percentage <20% AND clinical blood draw not planned.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 338 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2028-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yana Pikman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (15):
- United States (15):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital's and Clinics of Minnesota, Minneapolis, Minnesota
  - Washington University at St. Louis School of Medicine, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paolino J, Dimitrov B, Apsel Winger B, Sandoval-Perez A, Rangarajan AV, Ocasio-Martinez N, Tsai HK, Li Y, Robichaud AL, Khalid D, Hatton C, Gillani R, Polonen P, Dilig A, Gotti G, Kavanagh J, Adhav AA, Gow S, Tsai J, Li Y, Ebert BL, Van Allen EM, Bledsoe J, Kim AS, Tasian SK, Cooper SL, Cooper TM, Hijiya N, Sulis ML, Shukla NN, Magee JA, Mullighan CG, Burke MJ, Luskin MR, Mar BG, Jacobson MP, Harris MH, Stegmaier K, Place AE, Pikman Y. Integration of Genomic Sequencing Drives Therapeutic Targeting of PDGFRA in T-Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma. Clin Cancer Res. 2023 Nov 14;29(22):4613-4626. doi: 10.1158/1078-0432.CCR-22-2562. PMID 37725576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from August 17, 2016 to May 4, 2022.
Groups:
- Relapsed/Refractory Leukemia: Cohort 1: Relapsed/refractory leukemia
  * Acute lymphoblastic leukemia (ALL), first or greater relapse
  * Acute myeloid leukemia (AML), first or greater relapse
  * Leukemia refractory to induction chemotherapy
  * Other recurrent leukemia
  * Myelodysplastic syndrome (MDS), first or greater relapse, or refractory to initial therapy
- New Diagnosis: Cohort 2: New diagnosis
  * Acute myeloid leukemia (AML), new diagnosis (excluding acute promyelocytic leukemia (APL))
  * New diagnosis infant mixed-lineage leukemia (MLL)-rearranged ALL or low hypodiploid (<40 chromosomes) ALL
  * Rare leukemia- e.g., juvenile myelomonocytic leukemia (JMML), leukemia of ambiguous lineage
  * Secondary leukemia
  * Myelodysplastic syndrome (MDS) not eligible for stem cell transplant
Period: Overall Study
Arm/Group | Relapsed/Refractory Leukemia | New Diagnosis
Started | 236 | 102
Matched targeted therapy (MTT) data available | 157 | 74
Evaluable for primary endpoint | 101 | 0 (Only Cohort 1 is meant to address the primary outcome. Cohort 2 will be reported for secondary outcomes.)
Completed (A patient is completed if they completed the required follow-up and came off study.) | 14 | 9
Not Completed | 222 | 93
Not completed — Death | 94 | 14
Not completed — Lost to Follow-up | 4 | 1
Not completed — Subject withdrew consent | 1 | 0
Not completed — Unknown, data entry delayed | 123 | 78

BASELINE CHARACTERISTICS:
Population: This analysis dataset is comprised of all enrolled patients.
Groups:
- Relapsed/Refractory Leukemia: Cohort 1: Relapsed/refractory leukemia
  * Acute lymphoblastic leukemia (ALL), first or greater relapse
  * Acute myeloid leukemia (AML), first or greater relapse
  * Leukemia refractory to induction chemotherapy
  * Other recurrent leukemia
  * Myelodysplastic syndrome (MDS), first or greater relapse, or refractory to initial therapy
  After the screening procedures confirms patient eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Leukemia Profiling: Genetic profiling of leukemia cells will be performed and analyzed by an expert panel. Matched targeted therapy recommendation based on profiling results will be made if available. The recommendation, if available, will be communicated to the primary oncologist.
- New Diagnosis: Cohort 2: New diagnosis
  * Acute myeloid leukemia (AML), new diagnosis (excluding acute promyelocytic leukemia (APL))
  * New diagnosis infant mixed-lineage leukemia (MLL)-rearranged ALL or low hypodiploid (<40 chromosomes) ALL
  * Rare leukemia- e.g., juvenile myelomonocytic leukemia (JMML), leukemia of ambiguous lineage
  * Secondary leukemia
  * Myelodysplastic syndrome (MDS) not eligible for stem cell transplant
  After the screening procedures confirms eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Leukemia Profiling: Genetic profiling of leukemia cells will be performed and analyzed by an expert panel. Matched targeted therapy recommendation based on profiling results will be made if available. The recommendation, if available, will be communicated to the primary oncologist.
- Total: Total of all reporting groups
Arm/Group | Relapsed/Refractory Leukemia | New Diagnosis | Total
Number analyzed (Participants) | 236 | 102 | 338
Age, Continuous [Median (Full Range); unit: years] | 11.3 [0.5 to 28.7] | 10.2 [0.4 to 26.5] | 11.1 [0.4 to 28.7]
Age, Customized [Count of Participants; unit: Participants]
  Age (years) at sample: <1 years | 7 | 10 | 17
  Age (years) at sample: 1-9 years | 91 | 40 | 131
  Age (years) at sample: 10-17 years | 94 | 33 | 127
  Age (years) at sample: >=18 years | 44 | 19 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 51 | 164
  Male | 123 | 51 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 16 | 59
  Not Hispanic or Latino | 144 | 75 | 219
  Unknown or Not Reported | 49 | 11 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 9 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 14 | 33
  White | 127 | 60 | 187
  More than one race | 24 | 15 | 39
  Unknown or Not Reported | 51 | 4 | 55
Disease [Count of Participants; unit: Participants]
  AML | 89 | 70 | 159
  MDS | 4 | 2 | 6
  JMML | 2 | 2 | 4
  B-cell ALL | 111 | 1 | 112
  T-cell ALL | 14 | 2 | 16
  Infant MLL rearranged ALL | 2 | 4 | 6
  Leukemia of ambiguous lineage | 8 | 8 | 16
  Other rare leukemia | 2 | 4 | 6
  Secondary leukemia | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients With Actionable Alterations
Description: An actionable alteration was defined as a cancer-associated genomic event for which there was a targeted drug available. Actionable genetic alterations were identified by a combination of standard-of-care cytogenetics/fluorescence in situ hybridization (FISH) and sequencing performed as part of the study. This study is considered feasible if at least 13% of participants analyzed have profile data and identifiable actionable alterations. A 90% exact binomial confidence interval is presented for the rate of patients with actionable alterations to compare the observed rate against 13%.
Time Frame: Actionable alteration was identified based on a combination of fluorescence in situ hybridization (FISH)/cytogenetics and sequencing. Average time to full results was 2 weeks.
Population: The analysis dataset is comprised of the first 100 patients in Cohort 1, as defined per protocol. One patient in Cohort 2 was later identified to have relapsed/refractory disease, so therefore the analysis population contains 101 patients. The remainder of Cohort 1 patients and the entirety of Cohort 2 patients are represented in the analysis of secondary outcomes.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Relapsed/Refractory Leukemia: Cohort 1: Relapsed/refractory leukemia
  * Acute lymphoblastic leukemia, first or greater relapse
  * Acute myeloid leukemia, first or greater relapse
  * Leukemia refractory to induction chemotherapy
  * Other recurrent leukemia
  * Myelodysplastic syndrome (MDS), first or greater relapse, or refractory to initial therapy
  After the screening procedures confirms patient eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Leukemia Profiling: Genetic profiling of leukemia cells will be performed and analyzed by an expert panel. Matched targeted therapy recommendation based on profiling results will be made if available. The recommendation, if available, will be communicated to the primary oncologist.
- New Diagnosis: Cohort 2: New diagnosis
  * Acute myeloid leukemia, new diagnosis (excluding acute promyelocytic leukemia (APL))
  * New diagnosis infant MLL-rearranged ALL or low hypodiploid (<40 chromosomes) ALL
  * Rare leukemia- e.g., JMML, leukemia of ambiguous lineage
  * Secondary leukemia
  * Myelodysplastic syndrome (MDS) not eligible for stem cell transplant
  After the screening procedures confirms eligibility:
  * Leukemia Profiling will be performed
  * Identifying an actionable genomic alteration and making a matched targeted therapy treatment recommendation.
  Leukemia Profiling: Genetic profiling of leukemia cells will be performed and analyzed by an expert panel. Matched targeted therapy recommendation based on profiling results will be made if available. The recommendation, if available, will be communicated to the primary oncologist.
Arm/Group | Relapsed/Refractory Leukemia | New Diagnosis
Number analyzed (Participants) | 101 | 0
percentage of participants | 77 [69 to 84] |

2. Secondary Outcome: Rate of Somatic Genomic Alterations
Description: This Secondary Outcome will be addressed by describing the somatic genomic alterations in Cohort 1 (Relapsed/Refractory Leukemia arm) and Cohort 2 (New Diagnosis arm) that are discovered by genomic analyses.
Time Frame: 2 Years
Reporting Status: Not Posted, anticipated posting 2028-05

3. Secondary Outcome: Rate of Results Reporting
Description: This Secondary Outcome will be addressed by a description of the time of results reporting. Documentation of the time of sample receipt and processing, resources and personnel utilized at each step of the process, time to results reporting, interpretation and review by Expert panel and communication of results to the primary oncologist will be captured.
Time Frame: 2 Years
Reporting Status: Not Posted, anticipated posting 2028-05

4. Secondary Outcome: Parent's Feelings and Understanding of Genomic Testing
Description: This Secondary Outcome will be addressed by describing the hopes and concerns of parents of children with recurrent/refractory/high-risk de novo leukemia regarding genomic testing of their child's leukemia as well as their understanding of the testing and evaluate whether the hopes and concerns were realized following the return of results.
Time Frame: 2 Years
Reporting Status: Not Posted, anticipated posting 2028-05

5. Secondary Outcome: Analysis of Primary Leukemia Sensitivity Testing and Establishment of Xenograft Models
Description: This Secondary Outcome will be addressed by completing analysis of the primary leukemia sensitivity testing to a panel of drugs or shRNA and establishing xenograft models in dedicated participating research laboratories and conducting co-clinical trials with the recommended matched therapy once the animal model is established.
Time Frame: 2 Years
Reporting Status: Not Posted, anticipated posting 2028-05

ADVERSE EVENTS:
Time Frame: Adverse event data was not of interest or collected for this study since there was no treatment intervention involved. Mortality data was not monitored for the duration of study completion, and cause of death was not collected for patients for whom a status of death was provided by outside sites.
Description: Adverse event data was not of interest or collected for this study since there was no treatment intervention involved. Mortality data was not monitored for the duration of study completion, and cause of death was not collected for patients for whom a status of death was provided by outside sites.
Arm/Group | Relapsed/Refractory Leukemia | New Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT02670525/Prot_SAP_000.pdf